CLINICAL TRIAL: NCT03582735
Title: Effects of a Preoperative Neuromobilization Program Offered to Individuals With Carpal Tunnel Syndrome Awaiting Carpal Tunnel Release Surgery: a Pilot Randomized Controlled Trial
Brief Title: Preoperative Neuromobilization Exercises for Individuals With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Dany H. Gagnon, Senior researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DG_NM_15e; 2015-16-#19 (Other Grant/Funding Number: OPPQ and the Quebec Rehabilitation Research Network)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Ultrasound Imaging; Preoperative Care; Exercise Therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be allocated in two groups to receive either the experimental intervention (i.e., nerve gliding exercise program) or control intervention (i.e., no treatment)
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to participant allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve gliding exercise (Experimental): Three series of 15 daily repetition of the rehabilitation exercise targetting nerve excursion
  Interventions: Other: Nerve gliding exercise
- Control (No Intervention): No intervention according to current practice.

INTERVENTIONS:
Other: Nerve gliding exercise — A 4-week home-based nerve-gliding exercise program (NGEP) including isolated and coupled upper limb and neck movements. A specific mobilization was elaborated for each week of the program allowing to gradually increase the range of movement and inter-articular coordination.
  Arms: Nerve gliding exercise

SUMMARY:
Carpal tunnel syndrome is one of the major known disorders of the wrist and hand that causes pain, tingling sensations, weakness of the hand and functional limitations in daily tasks (for example: handling objects with the hands). In the early stages of the syndrome, some individuals may benefit from wearing wrist splint or cortisone infiltration. For those with ongoing symptoms, surgery is often indicated. However, some individuals may experience worsening of their condition while waiting for surgery. To aid those individuals, physiotherapists often recommend exercises that aim to "glide" the nerve inside the arm. Specifically, these exercises involve arm and neck movements in a specific order, with the aim of improving the motion of the median nerve in relation with its environment. These nerve gliding exercises may have a favorable effect on the median nerve and may improve pain and upper limb functional abilities. In this study, the investigators aim to evaluated the feasibility and effects of a preoperative nerve gliding exercises completed by individuals undergoing surgery

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome (CTS) is a common disorder characterized by alterations of the median nerve integrity at the carpal tunnel. The syndrome is classically recognized by chief complains of nocturnal or intermittent pain and paresthesia involving the median nerve sensory territory of the hand. In more severe condition, worsening of pain and paresthesia as well as thenar muscle atrophy may be present and lead to disability.

Many conservative treatments for CTS are available. Yet, the current literature only support the use of wrist splints and cortisone infiltration, which have been shown to provide only temporary relief for many individuals. Those with ongoing symptoms or severe conditions are often offered carpal tunnel decompression surgery. However, the costs related to the surgery and the increasing delays on waiting lists warrants the need for better conservative management. A preoperative rehabilitation exercise program based on nerve gliding exercise is advocated by physical therapists to manage physical impairments and functional limitations associated with CTS. These exercises can be implement at low cost in the setting of an home-based program.

The investigators aim to examine the feasibility and the efficacy of a preoperative home rehabilitation program based on nerve gliding exercises completed by individuals with carpal tunnel Syndrome waiting for decompression surgery.

In this trial, individuals awaiting carpal tunnel decompression surgery will be randomly allocated to either complete a preoperative nerve-gliding exercise program (experimental group) or no intervention (control group). Thirty participants confirmed with CTS by their attending hand surgeons and enlisted for carpal tunnel decompression will be recruited for this study conducted at the hospital of the Université de Montréal (CHUM), Montreal, Quebec, Canada. All individuals enrolled in the study will be prioritized on the surgical waiting list to receive their surgery five weeks after initiating the study in order to ensure consistency between different timeframes of the study.

The effects of the nerve-gliding exercise program will be assessed at baseline (T0) using standardized questionnaires, quantitative ultrasound measurements (including static and dynamic evaluations) of the median nerve, pinch grip strength and will be repeated after four weeks (T1; preoperative period) and four weeks following surgery (T2; postoperative period).

Feasibility metrics will be analyzed using descriptive statistics. A significant interaction between the group allocation (experimental vs. control) and time (T0 vs. T1 vs. T2) on the main outcomes will be evaluated using two-way mixed ANOVAs.

ELIGIBILITY:
Inclusion Criteria:

* EMG confirmed diagnosis of carpal tunnel syndrome
* Listed for carpal tunnel decompression

Exclusion Criteria:

* Previous trauma or surgery impairing motion of the upper limb
* Diabetes
* Thyroid disease
* Rheumatoid arthritis
* Recent pregnancy (< 3 months)
* Unable to communicate in English or French

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in different pain-related disabilities and cognitive-behavioral factors involved in the experience of pain measured by the West Haven-Yale Multidimensional Pain inventory (WHYMPI) | Baseline (T0), one month (T1), and two months (T2) following randomization
  The WHYMPI is comprised of 52 questions organized into subscales quantifying domains including two subscales specific to pain experience (i.e., pain interference (9 items), and pain severity (3 items)). Each question is rated on a Likert scale ranging from 0 to 6 and a mean score is computed for each subscale. A higher mean score represents higher disability (e.g., very intense pain or extreme interference). The French version of the WHYPMI has been adapted and validated and has demonstrated good repeatability (ICC > 0.75) when tested in adults with chronic musculoskeletal pain (Laliberté et al. 2008, Kerns, Turk, and Rudy 1985). The normalized minimal detectable change (MDC) for the WHYMPI for each of the five WHYMPI subscales range from MDC90%=15.4% (pain interference) to MDC90%=22.8% (emotional distress) (Bergström et al. 1999).
Change upper limb functional abilities measured with the Disability of the Arm, Shoulder and Hand (DASH) scale | Baseline (T0), one month (T1), and two months (T2) following randomization
  The DASH includes 30 questions covering participation and performance of daily activities with the upper limb as well as symptom severity in individuals with musculoskeletal upper limb disorder. Each question is rated on a Likert scale ranging from 1 to 5, where a higher weighted score (range 0-100) represents substantial functional limitations. The French version of the DASH has been adapted and validated and has demonstrated excellent repeatability (ICC = 0.91) when tested in adults with chronic musculoskeletal pain (Hudak, Amadio, and Bombardier 1996, Durand et al. 2005). The normalized MDC was established (MDC90% = 10.7%) (Greenslade et al. 2004).

SECONDARY OUTCOMES:
Change in median nerve cross sectional area at the carpal tunnel inlet measured by quantitative ultrasound imaging | Baseline (T0), one month (T1), and two months (T2) following randomization
  Static images of the median nerve's are acquired in the transverse plane at the level of the carpal tunnel inlet. The cross-sectional area of the median nerve is defined by semi-automatically outlining the inner border of the epineurium and will be assess offline using custom software. Median nerve cross-sectional area measurement has good repeatability ( > 0.88) when performed in asymptomatic adults. The normalized MDC was previously estimated for the cross-sectional area measurement (MDC90% = 6.2%)
Change in median nerve longitudinal excursion at the distal forearm measured by quantitative ultrasound imaging | Baseline (T0), one month (T1), and two months (T2) following randomization
  Cineloops of the median nerve are acquired during passive extension of the wrist using ultrasound imaging at the distal forearm. Three region of interest within the epineurium border are manually drawn and will be assess offline custom software. Median nerve longitudinal excursion has good repeatability ( > 0.84) when performed in a mixed population including asymptomatic individuals and individuals with carpal tunnel syndrome. The normalized MDC was previously estimated for the longitudinal excursion measurement (MDC90% = 34.1%)
Change in pinch grip strength | Baseline (T0), 4th week (T1), and four weeks following surgery (T2)
  Assessment of thumb strength (in kilogram) using hand held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Dany H Gagnon, PT, PhD, Principal Investigator — Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Locations (1):
- Centre Hospitalier Universitaire de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data that underlie the results submitted for publication in peer-reviewed journal (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement
URL: http://crir.ca